CLINICAL TRIAL: NCT02639026
Title: Phase I Trial Of Hypofractionated Radiotherapy In Combination With MEDI4736 And Tremelimumab For Patients With Metastatic Melanoma And Lung, Breast And Pancreatic Cancers
Brief Title: Trial Of Hypofractionated Radiotherapy In Combination With MEDI4736 And Tremelimumab For Patients With Metastatic Melanoma And Lung, Breast And Pancreatic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 23915
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Metastatic; Melanoma; Non Small Cell Lung Cancer (NSCLC); Breast Cancer; Pancreatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Pancreatic Neoplasms | interventions — Radiotherapy; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Subjects will receive 20 mg/kg MEDI4736 and 1 mg/kg tremelimumab in combination every 4 weeks for 4 doses, followed by 10 mg/kg MEDI4736 monotherapy every 2 weeks for 18 doses. The total duration of therapy is 12 months. Cohort 1 tests 8 Gy x 3 fractions
  Interventions: Radiation: Radiotherapy; Drug: MEDI4736; Drug: Tremelimumab
- Cohort 2 (Experimental): Subjects will receive 20 mg/kg MEDI4736 and 1 mg/kg tremelimumab in combination every 4 weeks for 4 doses, followed by 10 mg/kg MEDI4736 monotherapy every 2 weeks for 18 doses. The total duration of therapy is 12 months. Cohort 2 tests 17 Gy x 1 fraction.
  Interventions: Radiation: Radiotherapy; Drug: MEDI4736; Drug: Tremelimumab

INTERVENTIONS:
Radiation: Radiotherapy — two schedules of radiotherapy (8 Gy x 3 fractions and 17 Gy x 1 fraction)
Drug: MEDI4736 — 20 mg/kg MEDI4736 every 4 weeks for 4 doses, followed by 10 mg/kg MEDI4736 monotherapy every 2 weeks for 18 doses
Drug: Tremelimumab — 1 mg/kg every 4 weeks for 4 doses

SUMMARY:
The main purpose of this study is to determine how best to combine hypofractionated radiotherapy, MEDI4736, and tremelimumab and to determine how safe and tolerable hypofractionated radiotherapy, MEDI4736, and tremelimumab are when given together in subjects with metastatic, melanoma, non small cell lung cancer (NSCLC), breast cancer, and pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic melanoma,metastatic non-small cell lung cancer, metastatic breast cancer, or metastatic pancreatic adenocarcinoma relapsed or refractory to therapy as outlined below or patients with these malignancies who have declined, are or have become unable to tolerate (e.g. progressive chemotherapy-associated peripheral neuropathy), or were not eligible for standard therapy: Metastatic melanoma patients at any line of therapy, Metastatic non-small cell lung cancer patients who have relapsed or are refractory to at least one line of systemic anti-cancer therapy for metastatic disease, including cytotoxic chemotherapy or targeted therapy, Metastatic breast cancer patients who have relapsed or are refractory to at least one line of systemic anti-cancer therapy for metastatic disease, such as cytotoxic chemotherapy, hormonal therapy, or targeted therapy, Metastatic pancreatic adenocarcinoma who have relapsed or are refractory to at least one line of systemic anti-cancer therapy for metastatic disease, such as cytotoxic chemotherapy or targeted therapy
* At least two measurable lesions (including the index lesion) according to RECIST guidelines v1.1
* An index lesion measuring between 1cm - 7cm that is amenable to hypofractionated radiation therapy at the discretion of the treating radiation oncologist

  o Index lesions in the pancreas are excluded in the second cohort
* Age greater than or equal to 18 years
* Signed, written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate hematological function documented within 3 weeks prior to initial treatment based on: White blood cell ≥ 2,500 cells/ul without growth factor support, Absolute neutrophil count (ANC) ≥ 1,500 cells/ul without growth factor support, Hemoglobin ≥ 9 g/dL, Platelet count ≥ 100,000 platelets/ul, Adequate hepatic and renal function documented within 3 weeks prior to initial treatment based on: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN). For subjects with liver metastasis, ALT and AST ≤ 5 x ULN, Total bilirubin ≤1.5 x ULN except in patients with documented Gilbert's syndrome or liver metastasis, who must have a baseline total bilirubin ≤ 3.0 mg/dl, Serum creatinine ≤ 2.0 mg/dL
* Full recovery from the acute effects of prior cancer treatments, defined as effects having resolved to NCI CTCAE v4.03 Grade 0 or 1 with the exception of alopecia and certain laboratory values as listed above. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by MEDI4736 and tremelimumab may be included (eg, hearing loss, neuropathy) upon approval of the PI.
* For patients with central nervous system (CNS) metastases, metastases must be asymptomatic at the time of Day 1 of the study and meet the following criteria:
* At least 28 days without progression of CNS metastases as evidenced by magnetic resonance imaging (MRI) or computed tomography (CT) after last day of treatment with radiation to the CNS metastases
* At least 14 days since last dose of corticosteroids
* Must not have leptomeningeal disease or cord compression
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 180 days after the final dose of MEDI4736 and tremelimumab. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation for 180 days after the final dose of MEDI4736 and tremelimumab: Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are not post-menopausal (defined as 12 months with no menses with postmenopausal gonadotropin levels, luteinizing hormone [LH] and follicle-stimulating [FSH], or postmenopausal estradiol levels within the postmenopausal range according to local guidelines without an alternative medical cause), A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. The acceptable methods of contraception include barrier methods (male condom plus spermicide, Copper T intrauterine device, Levonorgesterel-releasing intrauterine system) or hormonal methods (implants, hormone shot or injection, combined pill, minipill, patch), Nonsterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception (as outlined above) from Day 1 through 90 days after receipt of the final dose of MEDI4736 and tremelimumab. In addition, they must refrain from sperm donation for 90 days after the final dose of investigational product.

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless in a follow-up period or the study is an observational or non-interventional study
* Prior treatment with anti-CTLA4, anti-PD-1, or anti-PD-L1 (approved or investigational agent)
* Concurrent treatment with any anticancer agent, including chemotherapy, immunotherapy, or biologic therapy. In breast cancer patients, concurrent use of hormonal therapy (but not trastuzumab) is acceptable provided hormonal therapy was initiated more than 30 days prior to treatment on this study.
* Treatment with any other investigational agent within 3 weeks prior to the first dose of DURVALUMAB (MEDI4736) and tremelimumab
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of DURVALUMAB (MEDI4736) and tremelimumab or still recovering from prior surgery Note: Local surgery of isolated lesions for palliative intent is acceptable
* Current or prior use of immunosuppressive medication within 14 days before the first dose of DURVALUMAB (MEDI4736) and tremelimumab with the exceptions of intranasal and inhaled corticosteroids, systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent, or steroids used transiently to control contrast agent allergies for radiographic studies.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone.
* History of sensitivity or allergy to monoclonal antibodies or immunoglobulin GActive infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Receipt of a live, attenuated vaccine within 30 days prior to the first dose of DURVALUMAB (MEDI4736) and tremelimumab Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Clinical contraindication to stereotactic body radiotherapy as determined by the investigator (e.g., active systemic sclerosis, active inflammatory bowel disease if bowel is within radiation field.)
* Prior radiotherapy that precludes the proposed treatment with hypofractionated radiotherapy
* Females who are pregnant, lactating, or intend to become pregnant during the participation of the study
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Other active invasive malignancy. History of non-invasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin, or ductal carcinoma in situ of the breast is allowed, as is history of other invasive malignancy that is in remission after treatment with curative intent.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. O'Hara, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States